CLINICAL TRIAL: NCT01176383
Title: A Protocol for an Randomised Controlled Trial of Smoking Cessation Success Rate With or Without a Genetic Test, "Respiragene", to Assess Lung Cancer Risk - an Exploratory Study
Brief Title: Impact of a Gene Test for Susceptibility to Lung Cancer in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sussex NHS Research Consortium (Other Government)
Collaborators: University of Surrey (Other); Lab 21, Cambridge (Unknown); NHS Research and Development (Other Government)
Responsible Party: Principal Investigator, John Nichols, Visiting Research fellow, University of Surrey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SPCRU1
Record Dates: First submitted 2010-08-03; First posted 2010-08-06 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Smoking Cessation
Keywords: Nicotine addiction; Behaviour; Gene test; Lung cancer; Lifetime risk of lung cancer in smokers
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Behavior; Lung Neoplasms | interventions — Risk Factors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): The control group will have a standard NHS cessation clinic experience
- Respiragene test and risk score (Experimental): Subjects will have a buccal swab taken at first attendance for a 12 gene test of SNP variants associated with risk of lung cancer. From the genetic data and clinical data (any history of COPD, family history of lung cancer in a first degree relative and age) a risk score is calculated from which a lifetime risk of lung cancer if the subject continues to smoke can be calculated. This is expected to be a powerful motivator to encourage smoking cessation.
  Interventions: Genetic: Respiragene test and risk score

INTERVENTIONS:
Genetic: Respiragene test and risk score — This 12 gene test used with other data (family history, age and spirometry result) to calculate lifetime risk of lung cancer in smokers who do not quit smoking. This intervention is expected to be a motivator to quit.
  Other Names: Respiragene test, Lab 21, Cambridge
  Arms: Respiragene test and risk score

SUMMARY:
Professor RP Young (Associate Professor of Medicine and Molecular Medicine, School of Biological Sciences, University of Auckland) and his team have developed a reliable genetic test "Respiragene" based on 20 single nucleotide polymorphisms that can be used (together with details of personal and family history) to calculate a smoker's lifetime risk of developing lung cancer. The expectation is that whatever the score (estimated lifetime risk will vary from 5% to 50%) the result will counter "optimism bias" of the smoker and encourage smoking cessation and this assumption is supported by previous research on similar tests and smoking cessation. The investigators plan to recruit two groups of subjects for smoking cessation but only one group will have the Respiragene test. Eight weekly smoking cessation sessions will be carried out at a Surrey primary care medical centre and will follow the usual format for National Health Service smoking cessation clinics using Champix (varenicline), counselling and the carbon monoxide breath meter but with added: evaluation questionnaires, fagerstrom nicotine addiction score, salivary cotinine (metabolite of nicotine) test. The main outcome measures will be estimation of smoking cessation at 4 weeks and six months after the completion of the seven smoking cessation sessions. Successful smoking cessation has to be confirmed by negative salivary cotinine at 4 weeks and six months and questionnaires will be used to estimate the influence of the Respiragene test compared with standard procedures such as counselling and the carbon monoxide breath readings.

DETAILED DESCRIPTION:
Despite the 5-10% probability of lung cancer in smokers, 50% do not believe they are at significantly increased risk Despite this, over 80% of smokers would like to know their personal risk of lung cancer. RP Young, a clinician at University of Auckland, has show a three way link between biomarkers for COPD, a set of 20 single nucleotide polymorphisms (SNPs) and lung cancer. He has demonstrated a strong correlation between a risk score (derived from family history of cancer, the 20 SNPs & clinical COPD) and the development of lung cancers whereas healthy smokers (who had not developed lung cancer) matched for age, gender and lifetime smoking habits had a relatively low risk score (n=446 lung cancer subjects, 484 healthy current smokers. The odds ratio for lung cancer risk varied from 0.2-3.2 depending on the genetic risk (p<0.001). The Auckland lung cancer risk score has a 90% sensitivity for a score of >4. The validity of 20 SNP gene test has also been confirmed in populations in Barcelona, Spain and Liverpool, United Kingdom. The test has been given the trade name "Respiragene".

Small uncontrolled trials of use of Respiragene in smoking cessation clinics in New Zealand and USA show an improvement in smoking cessation at six months after a Respiragene intervention with quit rates of 30-35%. The trial hypothesis is that smokers who have the Respiragene test and a full explanation of their risk score will have a better quit rate at 4 weeks and at six months (after completion of their eight weekly smoking cessation clinic sessions) than controls. Smoking cessation at the six month follow up will bw confirmed by testing for salivary cotinine. Based on data from Young's small trial, we also hypothesise that this uplift of quit rate will be seen for subjects with both high risk scores and average risk scores (there is no low risk category for smokers). These hypotheses are the basis of the primary end points.

The investigators will also be administering the same questionnaire to each subject and control twice, at 4 weeks and six months (after the smoking cessation course) that is primarily designed to evaluate the impact of the Respiragene test in relation to other influences:

* other components of the smoking cessation clinic sessions (salivary cotinine testing, carbon monoxide breath analyser, general clinic help and advice, clinic fact sheets)
* general environmental factors (cost of cigarettes, family pressure, work regulations, doctor's advice)

The results will be analysed using Statistical Package for the Social Sciences (SPSS) Statistics 17.0 computer programme.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-70 years
* Smoking more than 10 cigarettes daily

Exclusion Criteria:

* Aged under 20 years or over 70 years
* Smoking less than 10 cigarettes daily
* History of major depression and other psychiatric conditions, dementias and serious or terminal illness (cancers etc.).
* Patients on warfarin would be excluded due to interactions between warfarin and varenicline as varenicline will be used as the modern treatment of choice for smoking cessation.

Patients who did not wish to have a genetic test would be referred to the practice nurse for smoking cessation.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects versus controls who are non-smokers at 4 weeks and six months after completion of smoking cessation clinic | Nine months (from recruitment to completion)
  Subjects and controls will be reassessed at 4 weeks and six months after the last smoking cessation session to determine how many have genuinely stopped smoking. This will be confirmed at the six month follow up by measuring salivary cotinine to reveal any subjects who are being untruthful. The difference between quit rates in subjects and controls can then be calculated.

SECONDARY OUTCOMES:
Questionnaires to assess efficacy of Repiragene test as a motivator compared with other smoking cessation aids and motivators | Nine months (from recruitemnt to completion)
  All subjects will be asked to complete questionnaires (with assistance as needed) to assess the perceived value of the Respiragene test compared with other motivators (such as the price of cigarettes, family pressure etc.) and other motivational triggers used in the clinic (salivary cotinine, spirometry results etc.)

CONTACTS AND LOCATIONS:
Overall Officials: John Nichols, MB ChB, Principal Investigator — Surrey Primary Care Research Unit
Locations (1):
- The Integrated Care Partnership The Old Cottage Hospital Alexandra Road,, Epsom, Surrey, United Kingdom

REFERENCES:
- [Background] Young RP, Hopkins RJ, Hay BA, Epton MJ, Mills GD, Black PN, Gardner HD, Sullivan R, Gamble GD. Lung cancer susceptibility model based on age, family history and genetic variants. PLoS One. 2009;4(4):e5302. doi: 10.1371/journal.pone.0005302. Epub 2009 Apr 23. PMID 19390575
- [Background] Smith SM, Campbell NC, MacLeod U, Lee AJ, Raja A, Wyke S, Ziebland SB, Duff EM, Ritchie LD, Nicolson MC. Factors contributing to the time taken to consult with symptoms of lung cancer: a cross-sectional study. Thorax. 2009 Jun;64(6):523-31. doi: 10.1136/thx.2008.096560. Epub 2008 Dec 3. PMID 19052045
- [Background] Sanderson SC, O'Neill SC, White DB, Bepler G, Bastian L, Lipkus IM, McBride CM. Responses to online GSTM1 genetic test results among smokers related to patients with lung cancer: a pilot study. Cancer Epidemiol Biomarkers Prev. 2009 Jul;18(7):1953-61. doi: 10.1158/1055-9965.EPI-08-0620. Epub 2009 Jun 30. PMID 19567511
- [Background] Young RP, Hopkins R, Black PN, Eddy C, Wu L, Gamble GD, Mills GD, Garrett JE, Eaton TE, Rees MI. Functional variants of antioxidant genes in smokers with COPD and in those with normal lung function. Thorax. 2006 May;61(5):394-9. doi: 10.1136/thx.2005.048512. Epub 2006 Feb 7. PMID 16467073
- [Background] Young RP, Hopkins RJ, Christmas T, Black PN, Metcalf P, Gamble GD. COPD prevalence is increased in lung cancer, independent of age, sex and smoking history. Eur Respir J. 2009 Aug;34(2):380-6. doi: 10.1183/09031936.00144208. Epub 2009 Feb 5. PMID 19196816
- [Background] Young RP, Hopkins RJ, Hay BA, Epton MJ, Black PN, Gamble GD. Lung cancer gene associated with COPD: triple whammy or possible confounding effect? Eur Respir J. 2008 Nov;32(5):1158-64. doi: 10.1183/09031936.00093908. PMID 18978134
- [Background] Young RP, Hopkins RJ, Hay BA, Epton MJ, Mills GD, Black PN, Gardner HD, Sullivan R, Gamble GD. A gene-based risk score for lung cancer susceptibility in smokers and ex-smokers. Postgrad Med J. 2009 Oct;85(1008):515-24. doi: 10.1136/pgmj.2008.077107. PMID 19789190
- [Background] McBride CM, Bepler G, Lipkus IM, Lyna P, Samsa G, Albright J, Datta S, Rimer BK. Incorporating genetic susceptibility feedback into a smoking cessation program for African-American smokers with low income. Cancer Epidemiol Biomarkers Prev. 2002 Jun;11(6):521-8. PMID 12050092
- [Background] Sanderson SC, Humphries SE, Hubbart C, Hughes E, Jarvis MJ, Wardle J. Psychological and behavioural impact of genetic testing smokers for lung cancer risk: a phase II exploratory trial. J Health Psychol. 2008 May;13(4):481-94. doi: 10.1177/1359105308088519. PMID 18420756
- [Background] Parkes G, Greenhalgh T, Griffin M, Dent R. Effect on smoking quit rate of telling patients their lung age: the Step2quit randomised controlled trial. BMJ. 2008 Mar 15;336(7644):598-600. doi: 10.1136/bmj.39503.582396.25. Epub 2008 Mar 6. PMID 18326503
- [Background] Young RP, Hopkins RJ, Smith M, Hogarth DK. Smoking cessation: the potential role of risk assessment tools as motivational triggers. Postgrad Med J. 2010 Jan;86(1011):26-33; quiz 31-2. doi: 10.1136/pgmj.2009.084947. PMID 20065338
- [Background] Soulier-Parmeggiani L, Griscom S, Bongard O, Avvanzino R, Bounameaux H. One-year results of a smoking-cessation programme. Schweiz Med Wochenschr. 1999 Mar 13;129(10):395-8. PMID 10212973
- [Derived] Nichols JAA, Grob P, Kite W, Williams P, de Lusignan S. Using a genetic/clinical risk score to stop smoking (GeTSS): randomised controlled trial. BMC Res Notes. 2017 Oct 23;10(1):507. doi: 10.1186/s13104-017-2831-2. PMID 29061161
- [Derived] Nichols JA, Grob P, de Lusignan S, Kite W, Williams P. Genetic test to stop smoking (GeTSS) trial protocol: randomised controlled trial of a genetic test (Respiragene) and Auckland formula to assess lung cancer risk. BMC Pulm Med. 2014 May 1;14:77. doi: 10.1186/1471-2466-14-77. PMID 24884942